CLINICAL TRIAL: NCT00240669
Title: RESTIT : Evaluation of Resorbable Osteosynthesis Devices Versus Titanium in Maxillofacial Surgery - A Prospective Randomized Trial in Therapeutic Strategy
Brief Title: RESTIT : Evaluation of Resorbable Osteosynthesis Devices Versus Titanium in Maxillofacial Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004.366
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Maxillo-Facial Surgery
Keywords: Maxillo facial surgery,; osteosynthesis,; resorbable device

INTERVENTIONS:
Device: Resorbable device PLLA/PGA
Device: Titanium device

SUMMARY:
Primary objective : To evaluate the quality of fractures setting and osteotomy of the facial massif osteosynthesised with resorbable device PLLA/PGA compared with usual Titanium plates.

Secondary objective :

* To evaluate the resorbable device ergonomy versus Titanium.
* To evaluate the clinical tolerance of resorbable device versus Titanium.

Hypothesis :

Osteosynthesis with resorbable device demonstrates a non inferiority success probability regarding the success observed in osteosynthesis with Titanium, with a less important probability of re-operation.

Study duration : 14 months for each patient.

Study treatment :

* Group I : Resorbable device PLLA/PGA.
* Group II : Titanium device.

Study visits :

- Screening visit - Baseline with randomization and surgery - Day1 - Day 21 - Day 45(Traumatology)/Day 90 (orthognatic) - Month 6,12 and 14.

Randomization : Stratification by centres, mono or bimaxillar surgery and traumatologic or orthognatic criteria.

ELIGIBILITY:
Inclusion Criteria:

* 18<Age<50.
* One or more fractures of facial massif requiring a surgical setting with osteosynthesis plates.
* One or more osteotomy of facial massif requiring a surgical setting with osteosynthesis plates.
* Orally and written informed patient. Patient willing to participate the study.
* Signed informed consent.

Exclusion Criteria:

* Any previous surgery at the same operative site.
* Patient suffering from chronic affection which could interfere with bone consolidation.
* Corticotherapy, immunosuppressive or anticonvulsant treatment or long term antibiotherapy.
* Nursing or pregnant female.
* Patient with a high risk of non compliance to sudy visits.
* Unconscious patient.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 308
Dates: Start 2005-11

PRIMARY OUTCOMES:
The quality of fractures setting and osteotomy of the facial massif osteosynthesised with resorbable device PLLA/PGA will be evaluated by the notion of unperfect resuts.

SECONDARY OUTCOMES:
Evaluation of device ergonomy :
The operative time of each surgery will be monitored, to compare operative duration of operations ; the only variable will be the osteosynthesis method.
Clinical tolerance of the devices
pain (Visual Analogic Scale),
local inflammation,
scar disunion,
infection,
subcutaneous or submucous palpation of the plates.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BOULETREAU, MD, Principal Investigator — Hospices Civile de Lyon
Locations (1):
- Pierre Bouletreau, Lyon, France